CLINICAL TRIAL: NCT05146453
Title: Sternotomies and PectoIntercostal Fascia Blocks in Fast-Track Cardiac Anesthesiology
Acronym: SPIFFY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study published by different group; this study would not add to the existing knowledge.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114968
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Post-operative Pain
Keywords: sternotomy; regional anesthesia; pectointercoastal fascia block; fast-track cardiac surgery; post-operative pain; truncal nerve block; cardiac surgery; cardiac anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the physicians placing the nerve blocks will not be blinded to the treatment group. The post-operative care team including the nurses doing pain assessments and management will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group of patients will undergo placement of US guided pectointercostal fascia blocks.
  Interventions: Procedure: Pectointercostal fascia blocks
- Placebo (Placebo Comparator): The control group patients will receive the same intraoperative analgesia management. A PIF block will not be performed, instead, a peripheral nerve block catheter will be secured to the skin surface and connected to a CADD™ pump. As the catheter is taped to the skin surface the control group patients will not be exposed to the risks of peripheral nerve block placement.
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: Pectointercostal fascia blocks — PIF blocks will be placed at the conclusion of surgery with the surgical drapes in place. The blocks are performed using a high frequency linear transducer with aseptic technique. The ultrasound probe is placed longitudinally 3 cm from the sternum at the level of the 4th-6th intercostal space. Using an in-plane approach, an echogenic needle will be advanced into the fascial plane between pectoralis major and the external intercostal muscles. Peripheral nerve block catheters will then be inserted and secured to the skin surface with tegaderm. For patients weighing over 70 kg, 20 mL of 0.5% ropivacaine will be administered. This will be reduced to 15mL per side for patients weighing less than 70 kg. A CADD™ pump will be connected to each catheter and programmed to deliver 20 mL boluses of ropivacaine 0.2% starting at postoperative hour 2. The boluses will be staggered every 2 hours on alternate sides until hour 24. The catheters will be removed 24 hours post-operatively.
  Other Names: peripheral nerve block; regional anesthesia
  Arms: Intervention
Other: Placebo — The control group patients will receive the same intraoperative analgesia management. A PIF block will not be performed, instead, a peripheral nerve block catheter will be secured to the skin surface and connected to a CADD™ pump. As the catheter is taped to the skin surface the control group patients will not be exposed to the risks of peripheral nerve block placement.
  Arms: Placebo

SUMMARY:
This study is looking to see if a regional block placed on each side of the incision after surgery helps with pain relief. Ultrasound-guided pectointercostal fascia blocks will be placed at the conclusion of surgery following application of dressings. Patients will be in the supine position with the surgical drapes in place. The blocks are performed using a high frequency linear transducer with aseptic technique. The investigators hypothesize that placement of PIF blocks and catheters will decrease acute postoperative pain from midline sternotomy in fast track cardiac surgery patients compared to the current standard of care.

A physician will place an ultrasound guided pecto-intercostal fascial plane blocks bilaterally at the conclusion of surgery. They will also leave a catheter, similar to a small IV, between the muscle layers where the freezing medication goes. This will let the investigators give more freezing medication over the first 24 hours after surgery. The freezing medication blocks the pain signals from travelling to your brain from your incision, which might help participants need fewer narcotics after surgery.

Some of the research on this block shows a trend toward reduced pain, but the use of a catheter to allow repeat doses of freezing medication has not been studied. The investigators hope to show that this regional block means participants need less opioids (narcotics) in the first 2 days after their heart surgery.

In order to see whether the regional block is helpful there will be two groups of study participants. Both groups will receive infusion catheters covered with opaque bandages however one group will receive the study drug (ropivacaine) and the other will not (placebo). To reduce the risks to placebo group participants, those participants will have a catheter taped to their skin surface under an opaque dressing. This will give the illusion of block placement without the risks of a needle poking through skin. Both groups will still be given pain medications by IV or by mouth as needed after the surgery.

DETAILED DESCRIPTION:
Acute postoperative pain at median sternotomy sites is common in cardiac surgery patients. Inadequate control of acute pain can lead to sympathetic activation, hemodynamic sequelae, respiratory compromise, delirium and contributes to the development of chronic pain. Parental opioids have long been at the forefront of perioperative pain management for cardiac surgery patients, historically in large intravenous doses. With the onset of fast-track cardiac anesthesia (FTCA) which emphasizes reduced periods of post-operative mechanical ventilation, intensive care unit stay and overall health care cost; new strategies for managing post-operative pain in cardiac surgery patients are required. Opioid focused strategies contribute to many side effects including sedation, confusion, apnea, nausea, emesis, and ileusF , which can prevent effective fast tracking of these patients.

FTCA has highlighted the potential for regional anesthetic techniques to revolutionize post-operative cardiac surgery care. Though thoracic epidural analgesia offers excellent analgesia for post-sternotomy pain, the small but catastrophic risk of epidural hematoma in heparinized patients has hindered it from becoming standard of care. Over the last decade, various thoracic wall blocks have been developed and shown to benefit patients presenting for thoracic or breast surgeries, and sternotomies. Of these, fascial plane thoracic wall blocks offer the advantages of being simple to perform ultrasound equipment and having low complications rates.

One such block is the pectointercostal fascia (PIF) block which was first described in 2014 as an analgesic adjunct for breast procedures. In this block the fascial plane between the pectoralis major and internal intercostal muscles is infiltrated with local anesthetic with the aim of anesthetizing the anterior cutaneous branches of the intercostal nerves, thereby providing analgesia to the anterior chest wall from T2 to T6 with a single injection. The block can be placed with ultrasound guidance with the patient in the supine position - making it easy to place in the operating room or as a rescue block in CVICU. Despite the higher volumes of local anesthetic required for a plane block of this nature, previous studies have shown that the serum levels of local anesthetic remain well below the toxic rangeI,J. Injection into the fascial plane allows for excellent spread of local anesthetic along multiple rib spaces, precluding the need for multiple injections. It also opens up a space for placement of a catheter thus providing the option of longer term analgesia in postoperative patients. While PIF blocks avoid the hemodynamic side effects and risk of neuraxial complications associated with thoracic epidurals and paravertebral catheters they are not without risk. These risks include potential hemothorax, pneumothorax, chest wall hematoma, local anesthetic systemic toxicity and surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients presenting to the Mazankowski Heart Institute for operations via full midline sternotomy, i.e.: coronary artery bypass grafting, and/or single valve repair or single valve replacement who are expected to be fast track candidates post-operatively.
* patients scheduled for cardiac bypass grafting and/or single valve surgery requiring cardiopulmonary bypass.

Exclusion Criteria:

* Unstable or fluctuating cardiac condition (acute MI, HF, tamponade, type A dissection, ongoing refractory arrhythmia, LVEF <40%, massive transfusion protocol, reinstitution of CPB or other mechanical support)
* Alternative surgical approach (e.g. thoracotomy, mini sternotomy)
* Repeat sternotomy or emergency surgery
* Pregnancy or lactation
* Age <18
* Chronic pain
* Tolerance to opioids
* Active alcohol misuse disorder, IVDU or cannabis use >1g/d
* Allergy to local anesthetics
* Inability to provide informed consent
* High doses of steroids pre-operatively (>10 mg prednisone/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 12 hours
  Cumulative opioid consumption in milligrams of morphine in the first 12 hours after surgery.

SECONDARY OUTCOMES:
Opioid consumption in 24 hours | 24 hours post-operatively
  Amount of opioid consumed in 24 hours
Time to extubation | 24 hours
  Time until ETT is removed post-operatively.
Pain score | Every 6 hours for 24 hours post-operatively
  Pain score as reported using the numeric rating scale
ICU length of stay | 2 weeks
  Length of stay in ICU
Surgical site infection rate | 4 weeks
  Until hospital discharge
Local anesthetic systemic toxicity effects | 24 hours
  As evidenced by: tinnitus, perioral numbness, metallic taste

CONTACTS AND LOCATIONS:
Overall Officials: Wing Lam, Principal Investigator — University of Alberta
Locations (1):
- Gerhardus Heart van Rensburg, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelava M, Alfirevic A, Bustamante S, Hargrave J, Marciniak D. Regional Anesthesia in Cardiac Surgery: An Overview of Fascial Plane Chest Wall Blocks. Anesth Analg. 2020 Jul;131(1):127-135. doi: 10.1213/ANE.0000000000004682. PMID 32032103
- [Background] Fujii S, Bairagi R, Roche M, Zhou JR. Transversus Thoracis Muscle Plane Block. Biomed Res Int. 2019 Jul 7;2019:1716365. doi: 10.1155/2019/1716365. eCollection 2019. PMID 31360703
- [Background] Lloyd-Donald P, Lee WS, Hooper JW, Lee DK, Moore A, Chandra N, McCall P, Seevanayagam S, Matalanis G, Warrillow S, Weinberg L. Fast-track recovery program after cardiac surgery in a teaching hospital: a quality improvement initiative. BMC Res Notes. 2021 May 22;14(1):201. doi: 10.1186/s13104-021-05620-w. PMID 34022969
- [Background] Kar P, Ramachandran G. Pain relief following sternotomy in conventional cardiac surgery: A review of non neuraxial regional nerve blocks. Ann Card Anaesth. 2020 Apr-Jun;23(2):200-208. doi: 10.4103/aca.ACA_241_18. PMID 32275036
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Background] McDonald SB, Jacobsohn E, Kopacz DJ, Desphande S, Helman JD, Salinas F, Hall RA. Parasternal block and local anesthetic infiltration with levobupivacaine after cardiac surgery with desflurane: the effect on postoperative pain, pulmonary function, and tracheal extubation times. Anesth Analg. 2005 Jan;100(1):25-32. doi: 10.1213/01.ANE.0000139652.84897.BD. PMID 15616047
- [Background] Nasr DA, Abdelhamid HM, Mohsen M, Aly AH. The analgesic efficacy of continuous presternal bupivacaine infusion through a single catheter after cardiac surgery. Ann Card Anaesth. 2015 Jan-Mar;18(1):15-20. doi: 10.4103/0971-9784.148314. PMID 25566704
- [Background] Lee CY, Robinson DA, Johnson CA Jr, Zhang Y, Wong J, Joshi DJ, Wu TT, Knight PA. A Randomized Controlled Trial of Liposomal Bupivacaine Parasternal Intercostal Block for Sternotomy. Ann Thorac Surg. 2019 Jan;107(1):128-134. doi: 10.1016/j.athoracsur.2018.06.081. Epub 2018 Aug 28. PMID 30170012
- [Background] Chin KJ, Versyck B, Pawa A. Ultrasound-guided fascial plane blocks of the chest wall: a state-of-the-art review. Anaesthesia. 2021 Jan;76 Suppl 1:110-126. doi: 10.1111/anae.15276. PMID 33426660
- [Background] Nielsen S, Degenhardt L, Hoban B, Gisev N. A synthesis of oral morphine equivalents (OME) for opioid utilisation studies. Pharmacoepidemiol Drug Saf. 2016 Jun;25(6):733-7. doi: 10.1002/pds.3945. Epub 2015 Dec 22. PMID 26693665